CLINICAL TRIAL: NCT00789230
Title: Mesh Versus Suture Repair for Umbilical Hernias: a Double Blinded, Randomised Controlled Clinical Trial
Brief Title: Mesh Versus Suture Repair for Umbilical Hernias
Acronym: HUMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruth Kaufmann, MD (Other)
Responsible Party: Sponsor-Investigator, Ruth Kaufmann, MD, R. Kaufmann, Erasmus Medical Center
Organization: Erasmus Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HUMP
Record Dates: First submitted 2008-11-09; First posted 2008-11-11 (Estimated); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Umbilical Hernia
Keywords: umbilical; hernia; mesh
MeSH Terms: conditions — Hernia, Umbilical; Hernia

STUDY DESIGN:
Intervention Model Description: Suture versus mesh repair in umbilical hernia patients
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- primary suture (Active Comparator)
  Interventions: Procedure: primary suture closure
- mesh enforced closure (Active Comparator)
  Interventions: Device: mesh enforced closure

INTERVENTIONS:
Procedure: primary suture closure — primary suture closure of hernia
  Arms: primary suture
Device: mesh enforced closure — mesh enforced closure of hernia
  Arms: mesh enforced closure

SUMMARY:
The purpose of the present study is to investigate whether or not the use of mesh is indicated in the repair of all size umbilical hernias as to reduce the rate of recurrence. This method is regularly used in umbilical hernia reconstruction although most surgeons repair small hernias using suture repair (fascia adaptation). Especially risk factors for hernia recurrence such as hernia size and BMI > 30 kg/m2 need to be evaluated and correlated to the method of hernia repair.

DETAILED DESCRIPTION:
Purpose The purpose of the present study is to investigate whether or not the use of mesh is indicated in the repair of all size umbilical hernias as to reduce the rate of recurrence. This method is regularly used in umbilical hernia reconstruction although most surgeons repair small hernias using suture repair (fascia adaptation). Especially risk factors for hernia recurrence such as hernia size and BMI > 30 kg/m2 need to be evaluated and correlated to the method of hernia repair.

Study design Randomised controlled, double blinded, multi-centre trial. 300 consecutive patients with an umbilical hernia will be included in the study. Patients will be randomised in one of two groups of 150 patients each. Group 1 will include patients that will undergo primary (suture) repair; group 2 umbilical hernias will be repaired using a pre-peritoneal, flat polypropylene mesh in a tension free fashion.

Stratification will be utilized for the size of the hernia (1-2 cm or ≥2-4 cm) and the participating centre. Patients will visit the outpatient clinic after 2-3 weeks and after 3, 12 and 24 months.

The cumulative hernia recurrence rate during the 2-years follow-up period will be the primary outcome of the study. Complications, pain and QOL are secondary endpoints.

Statistical analysis All analyses will be performed according to the intention to treat principle and as specified in the protocol.

Financial support None.

ELIGIBILITY:
Inclusion Criteria:

* Primary umbilical hernia
* Signed Informed consent

Exclusion Criteria:

* Umbilical hernia ≥ 4 cm diameter
* Recurrence
* Midline laparotomy
* Ascites/Cirrhosis
* ASA score IV or above
* Incarcerated hernia/emergency procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2006-01; Primary Completion 2015-04 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
hernia recurrence rate | 24 months

SECONDARY OUTCOMES:
Post-operative morbidity and complications | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: J. Jeekel, MD, PhD, Principal Investigator — Erasmus Medical Center; J.F. Lange, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (12):
- Germany (2):
  - Studienzentrum der Deutschen Gesellschaft für Chirurgie, Heidelberg
  - University of Witten/Herdecke, Witten
- Multimedica, Milan, Italy
- Netherlands (9):
  - Erasmus University Medical Center, Rotterdam, South Holland
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Wilhelmina Ziekenhuis, Assen
  - Reinier de Graaf Gasthuis, Delft
  - Havenziekenhuis, Rotterdam
  - Ikazia, Rotterdam
  - Maasstad Ziekenhuis, Rotterdam
  - Máxima Medisch Centrum, Veldhoven
  - Isala, Zwolle

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kaufmann R, Halm JA, Eker HH, Klitsie PJ, Nieuwenhuizen J, van Geldere D, Simons MP, van der Harst E, van 't Riet M, van der Holt B, Kleinrensink GJ, Jeekel J, Lange JF. Mesh versus suture repair of umbilical hernia in adults: a randomised, double-blind, controlled, multicentre trial. Lancet. 2018 Mar 3;391(10123):860-869. doi: 10.1016/S0140-6736(18)30298-8. Epub 2018 Feb 17. PMID 29459021